CLINICAL TRIAL: NCT05456113
Title: Cannabidiol and Vascular Reactivity to Skin Sensory Nerve Stimulation
Brief Title: Topical Cannabidiol Application and Skin Vascular Reactivity
Acronym: cannabidiol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Lacy Alexander, Professor of Kinesiology, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20515
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Vehicle control, does not contain cannabidiol
  Interventions: Biological: Cannabidiol
- Cannabidiol (Experimental): Active ingredient experimental arm, contains full spectrum connabidiol
  Interventions: Biological: Cannabidiol

INTERVENTIONS:
Biological: Cannabidiol — Urbal Activ Extra Strength CBD Body Strong Balm applied to region of forearm to be stimulated by iontophoresis machine

SUMMARY:
Cannabidiol, or CBD, is an over-the-counter "nutraceutical" that is more commonly being used by healthy adults for pain management, recovery from strenuous exercise, and general wellness. However, little research exists on the effects of CBD in otherwise healthy individuals. This study uses iontophoresis, a common technique used in physical therapy, to determine the effectiveness of topical CBD in lessening the reflex increased cutaneous vascular conductance response to stimulation of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older
* English speaking
* Non-obese class III, BMI ≤ 39.9
* Normal HbA1C of <6.5%

Exclusion Criteria:

* Abnormal resting heart rate (<60 or >100 bpm) or BP (systolic <100 or >129 mmHg, diastolic <60 or >100 mmHg) values
* Rash, skin disease, disorders of pigmentation
* Known skin allergies
* Diabetes
* Nicotine use (e.g. smoking, chewing tobacco, vaping, etc.)
* Illegal drug use
* Recent (within the last 30 days) CBD users either topical or oral
* Allergy or hypersensitivity to investigational agents
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Cutaneous Vascular Conductance | ~5 hours
  pulse units as measured by laser Doppler flowmetry

CONTACTS AND LOCATIONS:
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States